## **Consent Form for Participants Able to Give Consent**

V1.0, 20 March 2024
Centre name: University College of Osteopathy, London, UK
Study Protocol number: N/A

Full Title of Project: A Multimodal Manual Therapy-Based Intervention for People with Painful

Diabetic Neuropathy: Feasibility of a Randomised Controlled Trial (NeuOst)

Name of Principal Investigator: Dr David Hohenschurz-Schmidt

Contact details:

Phone: 07523629286

Email: David.Schmidt@uco.ac.uk

Postal: University College of Osteopathy

275 Borough High Street London SE1 1JE, UK

Please initial boxes to indicate your consent to individual items.

1. I confirm that I have read and understand the participant information sheet version 1.0 dated 20 March 2024 for the research project titled 'NeuOst: A Multimodal Manual Therapy-Based Intervention for People with Painful Diabetic Neuropathy: Feasibility of a Randomised Controlled Efficacy Trial' and have had the opportunity to ask questions which have been answered to my satisfaction. 2. (Consent required for participation.) 3. I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. (Required for participation.) 4. I understand that sections of any of my medical notes may be looked at by responsible individuals from University College of Osteopathy, London, or from regulatory authorities where it is relevant to my taking part in this research. (Required for participation.) 5. I understand that data collected from me are a gift donated to University College of Osteopathy and that I will not personally benefit financially if this research leads to an invention and/or the successful development of a new test, medication treatment, product or service. (Required for participation.) 6. I consent to the open sharing of any data collected during this trial that cannot be traced back to me. (Required for participation.) 7. I consent to take part in the research project titled 'NeuOst: A Multimodal Manual Therapy-Based Intervention for People with Painful Diabetic Neuropathy: Feasibility of a Randomised Controlled Efficacy Trial'. (Required for participation.)

| th or in the developm<br>an academic institutions<br>se outside of the Uni | collected from me to be<br>nent of a new test, med<br>on or commercial comp<br>ted Kingdom (which | dical |
|---|---|---|
| th or in the developm<br>an academic institutions<br>se outside of the Uni | nent of a new test, med<br>on or commercial comp<br>ted Kingdom (which | dical |
| | ed will keep this inform agree.) | ation |
| rposes. | | corded |
| on to the treating oste | eopath) for quality assu | |
| interviews with the | research team about n | ny |
| | | in any |
| he collection of infor | mation about serious h | nealth-related events, |
| mary of the study re | sults. | |
| Signature | Date | |
| | atment sessions being poses. Attial the box if you attend sessions being on to the treating oster into the treating oster interviews with the contacted at the end interviews with the contacted about the posterior study. (Optional withdraw your consense collection of informect for several month.) | atment sessions being observed by medical on to the treating osteopath) for quality assumitial the box if you agree.) contacted at the end of the study about the interviews with the research team about not study. (Optional item. Only initial the contacted about the possibility to take part initial the box if you agree.) withdraw your consent for data collection a the collection of information about serious he ect for several months after study initiation many of the study results. |

1 copy for participant; 1 copy for Principal Investigator; 1 copy for clinical notes

To ensure confidence in the process and minimise risk of loss, all consent forms <u>must</u> be printed, presented, and stored in double sided format.